CLINICAL TRIAL: NCT01627704
Title: 16α-[18F]-Fluoro-œstradiol PET: an in Vivo Biomarker Predicting Response to Hormone Treatment of Metastatic Breast Cancer?
Brief Title: Fluoroestradiol PET Imaging in Predicting Response to Hormone Therapy of Breast Cancer
Acronym: ESTROTEPREDIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P110113; IDRCB (Other: 2011/005043-27)
Record Dates: First submitted 2012-06-14; First posted 2012-06-26 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Metastatic Breast Cancer
Keywords: PET/CT,fluoroestradiol (18F); breast cancer; metastatic; prediction of response; hormone therapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluoroestradiol (18F) (Other)
  Interventions: Drug: Fluoroestradiol (18F)

INTERVENTIONS:
Drug: Fluoroestradiol (18F) — 2-4 MBq/kg body mass, one single IV injection

SUMMARY:
Compare the response rate after 6 months of hormone treatment (or a major change in hormone treatment) in metastatic breast cancer, according to the uptake of FES in metastatic lesions taking-up FDG on PET/CT at baseline. Hypothesis: best response rate will be observed in patients with all metastases taking up FES prior to treatment.

DETAILED DESCRIPTION:
Main objective: Compare the response rate after 6 months of hormone treatment (or a major change in hormone treatment) in metastatic breast cancer, according to the uptake of FES in metastatic lesions taking-up FDG on PET/CT at baseline.

Secondary objectives:

* evaluate diagnostic performance of FES PET/CT
* determine whether FES PET/CT is able to detect metastases that are not visible on FDG PET/CT. This point may constitute a direct benefit for the patient
* precise the nature of discordant FES/FDG foci
* validate and improve the interpretation criteria for FES PET/CT
* confirm the perfect tolerance

ELIGIBILITY:
Inclusion Criteria:

* Post menopausal
* age > 17
* WHO 0-2
* Metastatic adenocarcinoma of the breast
* Treated by antihormone treatment during around 5 years withdrawn for at least 3 months OR metastatic cancer at diagnosis having received no more than one line of hormone treatment
* Life expectancy > 6 months
* Hormone-dependent cancer initially demonstrated by hormone receptors in the tumour
* Presence of oestrogen receptors proven with immunohistochemistry (> 10%) and HER2 determined by immunohistochemistry or FISH (on primary tumour or a metastasis)
* Metastatic recurrence on FDG PET dating less than 1 month, confirmed by another modality (contrast-enhanced CT, MRI, ultrasonography, bone scintigraphy or PET/CT, other)
* FDG PET/CT available on PACS or CD DICOM III format 11
* Informed consent obtained

Exclusion Criteria:

* Other evolutive malignant disease or acute or chronic infectious disease
* Chemotherapy during the last 3 months or change in treatment since FDG PET/CT.
* Isolated liver metastasis (high FES uptake by normal liver)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Response rate six months after induction or major change in hormone therapy for metastatic breast cancer. | at 6 months
  Response rate six months after induction or major change in hormone therapy for metastatic breast cancer. Response will be determined according to RECIST 1.1 criteria for each patient.

SECONDARY OUTCOMES:
Number of visible non-physiologic foci on FES PET and on the corresponding FDG PET, during centralised reading sessions by masked readers. | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Khaldoun KERROU, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Médecine Nucléaire, Hôpital Tenon, Paris, France